CLINICAL TRIAL: NCT00215644
Title: Randomized Phase II Open-Label Controlled Study of EMD 72000 (Matuzumab), in Combination With the Chemotherapy Regimen ECX or the Chemotherapy Regimen ECX Alone as First-line Treatment in Subjects With Metastatic Esophago-Gastric Adenocarcinoma
Brief Title: Matuzumab Treatment With Epirubicin, Cisplatin and Capecitabine (ECX) in Esophago-Gastric Cancer
Acronym: MATRIX EG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD 72000-032; 2005-000146-36 (EudraCT Number)
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Esophagus; Gastric; Adenocarcinoma; EGFR; matuzumab; EMD 72000; randomized; Epirubicin; cisplatin; capecitabine; Metastatic Esophago-Gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma | interventions — matuzumab; Epirubicin; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab (Experimental)
  Interventions: Drug: Matuzumab; Drug: Epirubicin; Drug: Cisplatin; Drug: Capecitabine
- ECX Only (Active Comparator)
  Interventions: Drug: Epirubicin; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Matuzumab — Participants will receive matuzumab 800 milligrams (mg) intravenously (IV) every week, until disease progression (PD), unacceptable toxicity, death, or consent is withdrawn.
  Other Names: EMD 72000
  Arms: Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab
Drug: Epirubicin — Participants will receive epirubicin 50 milligrams per square meter (mg/m^2) on Day 1 of 21-day cycle up to a maximum of 8 cycles.
Drug: Cisplatin — Participants will receive cisplatin 60 mg/m^2 on Day 1 of 21-day cycle up to a maximum of 8 cycles.
Drug: Capecitabine — Participants will receive capecitabine 1250 mg/m^2 daily in a 21-day cycles up to a maximum of 8 cycles.

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of experimental treatment matuzumab and ECX chemotherapy, with ECX chemotherapy. Participants invited to take part have metastatic cancer of the esophagus (gullet) or stomach.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric adenocarcinoma or adenocarcinoma of the lower third of the esophagus
* Metastatic disease
* Immunohistological evidence of Epidermal Growth Factor Receptor (EGFR) expression from archived tissues
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1
* At least 1 measurable lesion (modified World Health Organization criteria)

Exclusion Criteria:

* Previous chemotherapy, unless neo-adjuvant or adjuvant therapy completed greater than (>) 12 months prior to study treatment
* Radiotherapy or major surgery within 4 weeks prior to treatment
* Brain metastases
* Peripheral neuropathy or ototoxicity greater than or equal to (>/=) Grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events Version 3 [NCICTC V3])
* Abnormal electrocardiogram (ECG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-08-31 (Actual); Primary Completion 2008-07-31 (Actual); Study Completion 2008-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (22):
- Germany (4):
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Oldenburg
  - Research Site, Recklinghausen
- Spain (4):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Valencia
- Switzerland (4):
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Sankt Gallen
- United Kingdom (10):
  - Research Site, Northwood, Middlesex
  - Research Site, Bournemouth
  - Research Site, Cambridge
  - Research Site, Chelmsford
  - Research Site, Guildford
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Northwood
  - Research Site, Portsmouth

REFERENCES:
- [Result] Rao S, Starling N, Cunningham D, Sumpter K, Gilligan D, Ruhstaller T, Valladares-Ayerbes M, Wilke H, Archer C, Kurek R, Beadman C, Oates J. Matuzumab plus epirubicin, cisplatin and capecitabine (ECX) compared with epirubicin, cisplatin and capecitabine alone as first-line treatment in patients with advanced oesophago-gastric cancer: a randomised, multicentre open-label phase II study. Ann Oncol. 2010 Nov;21(11):2213-2219. doi: 10.1093/annonc/mdq247. Epub 2010 May 23. PMID 20497967

RESULTS

PARTICIPANT FLOW:
Groups:
- Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab: Participants received matuzumab 800 mg IV every week and epirubicin 50 mg/m^2, cisplatin 60 mg/m^2 on Day 1 and capecitabine 1250 mg/m^2 daily in a 21-day cycles (ECX). A maximum of 8 cycles of ECX were administered and after 8 cycles, matuzumab alone was continued until PD, unacceptable toxicity, death, or consent was withdrawn. An observation period of at least 1 hour was specified between the end of the matuzumab infusion and the start of epirubicin administration when these treatments were given on the same day.
- ECX Only: Participants received epirubicin 50 mg/m^2, cisplatin 60 mg/m^2 on Day 1 and capecitabine 1250 mg/m^2 daily in a 21-day cycles (ECX). A maximum of 8 cycles of ECX were administered unless there was evidence of PD, or unacceptable toxicity, death occurred or consent was withdrawn.
Period: Overall Study
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Started | 36 | 36
Treated | 35 | 36
Completed | 0 | 0
Not Completed | 36 | 36
Not completed — Disease Progression | 28 | 10
Not completed — Adverse Event | 2 | 9
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 3 | 15
Not completed — Randomized but Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who received at least 1 cycle of matuzumab or any component of ECX.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Median (Full Range); unit: years] | 59 [29 to 79] | 64 [36 to 76] | 62 [29 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Assessed by Independent Review Committee
Description: Objective response was defined as having a complete response (CR) or a partial response (PR). Response assessment was performed using modified World Health Organization (WHO) criteria. CR: disappearance of all index and non-index lesions, without appearance of any new lesion. PR: greater than (>) 50 percent (%) decrease from baseline in sum of product of diameters of index lesions, without appearance of any new lesion.
Time Frame: Baseline up to PD or death due to any cause (up to approximately 3 years)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Number analyzed (Participants) | 35 | 36
percentage of participants | 31 [17 to 49] | 58 [41 to 74]

2. Secondary Outcome: Duration of Objective Response Assessed by Independent Review Committee
Description: Objective response was defined as having a CR or a PR. Response assessment was performed using modified WHO criteria. CR: disappearance of all index and non-index lesions, without appearance of any new lesion. PR: >50% decrease from baseline in sum of product of diameters of index lesions, without appearance of any new lesion. Duration of objective response was defined as time from first appearance of CR or PR to time of PD (PD: >25% increase in one or more lesions, or appearance new lesions) or death. Duration of objective response was to be assessed using Kaplan-Meier analysis.
Time Frame: From first documented objective response to PD or death due to any cause (up to approximately 3 years)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Number analyzed (Participants) | 35 | 36
months | NA [NA to NA] — Data could not be estimated because less than 50% of participants were reported with objective response. | NA [NA to NA] — Data could not be estimated because less than 50% of participants were reported with objective response.

3. Secondary Outcome: Progression-Free Survival
Description: PFS was defined as the time from randomization to the first documentation of PD or to death due to any cause, whichever occurred first. PD: >25% increase in one or more lesions, or appearance new lesions. PFS was estimated using Kaplan-Meier analysis.
Time Frame: Baseline up to PD or death due to any cause (up to approximately 3 years)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Number analyzed (Participants) | 35 | 36
months | 4.8 [2.9 to 8.1] | 7.1 [4.4 to 8.5]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from randomization to death (due to any cause). OS was estimated using Kaplan-Meier analysis.
Time Frame: Baseline until death due to any cause (up to approximately 3 years)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Number analyzed (Participants) | 35 | 36
months | 9.4 [7.5 to 16.2] | 12.2 [9.8 to 13.8]

5. Secondary Outcome: Best Overall Change From Baseline in European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (GHS)/Quality of Life (QoL) Score
Description: EORTC QLQ-C30 included GHS/QoL, functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Most questions from EORTC QLQ-C30 were a 4-point scale (1/Not at All to 4/Very Much), except Items 29-30, which comprise GHS scale and were a 7-point scale (1/Very Poor to 7/Excellent). For this instrument, GHS/QOL was linearly transformed and ranged 0-100, where lower scores indicate poorer functioning (e.g., worsening) and higher scores indicate better functioning (e.g., improvement). EORTC QLQ-C30 GHS/QoL score at baseline and best overall change from baseline (throughout study) are reported.
Time Frame: Baseline (Day 1), Post Baseline (Up to 3 Years)
Population: ITT population. Here, overall number of participants analyzed = participants who were evaluable for this outcome and "Number analyzed" = participants evaluable for specified timepoint for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Number analyzed (Participants) | 30 | 33
units on a scale
  Baseline | 53.3 (27.3) | 67.9 (22.4)
  Post-Baseline: number analyzed (Participants) | 21 | 32
  Post-Baseline | 0.0 (28.1) | -10.0 (33.9)

6. Secondary Outcome: Protein Biomarkers Levels
Time Frame: Baseline up to approximately 3 years
Population: Data for this outcome was not collected from any of the participant; hence, no data available for reporting.
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With Anti-Matuzumab Antibodies
Time Frame: Baseline up to approximately 3 years
Population: Data for this outcome was not collected from any of the participant; hence, no data available for reporting.
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Matuzumab Serum Concentration
Time Frame: Baseline up to approximately 3 years
Population: Data for this outcome was not collected from any of the participant; hence, no data available for reporting.
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Only selected AEs were collected and reported.
Arm/Group | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab | ECX Only
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 35/35 | 36/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epirubicin, Cisplatin, Capecitabine (ECX)+Matuzumab (N=35) | ECX Only (N=36)
Neutropenia (Blood and lymphatic system disorders) | 13 | 12
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Fatigue/lethargy (General disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Skin disorders (Skin and subcutaneous tissue disorders) | 23 | 11
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Palmar plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 2 | 3
Pulmonary embolism (Vascular disorders) | 3 | 1
Infection (Infections and infestations) | 1 | 2
Hypokalaemia (Investigations) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No